CLINICAL TRIAL: NCT02202772
Title: A Phase I/II Trial for the Use of Intravesical Cabazitaxel, Gemcitabine, and Cisplatin (CGC) in the Treatment of BCG-Refractory Non-muscle Invasive Urothelial Carcinoma of the Bladder Cancer
Brief Title: Intravesical Cabazitaxel, Gemcitabine, and Cisplatin (CGC) in the Treatment Urothelial Carcinoma of the Bladder
Acronym: CGC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guarionex J. Decastro (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Guarionex J. Decastro, Associate Professor of Urology at the Columbia University Medical, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAM8506
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma of the Urinary Bladder
Keywords: Urothelial; Cisplatin; Gemcitabine; Cabazitaxel; Bladder; Carcinoma; Bacillus Calmette-Guerin; Intravesical; Recurrent; Non-muscle; Invasive; Cancer
MeSH Terms: conditions — Carcinoma; Recurrence; Neoplasms | interventions — cabazitaxel; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Gem and Low Cab (Experimental): Gemcitabine: Intravesical; 2000mg/100ml; 1 time a week for 6 weeks; 2 hours Cabazitaxel: Intravesical; 2.5mg/100ml; 1 time a week for 6 weeks; 2 hours
  Interventions: Drug: Cabazitaxel; Drug: Gemcitabine
- Gem and High Cab (Experimental): Gemcitabine: Intravesical; 2000mg/100ml; 1 time a week for 6 weeks; 2 hours Cabazitaxel: Intravesical; 5mg/100ml; 1 time a week for 6 weeks; 2 hours
  Interventions: Drug: Cabazitaxel; Drug: Gemcitabine
- Gem, High Cab, and Low Cis (Experimental): Gemcitabine: Intravesical; 2000mg/100ml; 1 time a week for 6 weeks; 2 hours Cabazitaxel: Intravesical; 5mg/100ml; 1 time a week for 6 weeks; 2 hours Cisplatin: Intravesical; 66mg/100ml; 1 time a week for 6 weeks; 2 hours
  Interventions: Drug: Cabazitaxel; Drug: Gemcitabine; Drug: Cisplatin
- Gem, High Cab, Mod Cis (Experimental): Gemcitabine: Intravesical; 2000mg/100ml; 1 time a week for 6 weeks; 2 hours Cabazitaxel: Intravesical; 5mg/100ml; 1 time a week for 6 weeks; 2 hours Cisplatin: Intravesical; 80mg/100ml; 1 time a week for 6 weeks; 2 hours
  Interventions: Drug: Cabazitaxel; Drug: Gemcitabine; Drug: Cisplatin
- Gem, High Cab, High Cis (Experimental): Gemcitabine: Intravesical; 2000mg/100ml; 1 time a week for 6 weeks; 2 hours Cabazitaxel: Intravesical; 5mg/100ml; 1 time a week for 6 weeks; 2 hours Cisplatin: Intravesical; 100mg/100ml; 1 time a week for 6 weeks; 2 hours
  Interventions: Drug: Cabazitaxel; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Cabazitaxel — Intravesical instillation of the Cabazitaxel for 2 hours
  Other Names: Jevtana
Drug: Gemcitabine — Intravesical instillation of Gemcitabine for 2 hours
  Other Names: Gemzar
Drug: Cisplatin — Intravesical installation of Cisplatin for 2hours
  Other Names: Platinol, Platinol-AQ
  Arms: Gem, High Cab, High Cis; Gem, High Cab, Mod Cis; Gem, High Cab, and Low Cis

SUMMARY:
The investigators intend to evaluate the safety and toxicity proﬁle of intravesically administered multidrug regimen of Cabazitaxel, Cisplatin and Gemcitabine in treatment refractory Transitional Cell Carcinoma.The investigators propose to conduct a combined phase I trial to assess the safety, toxicity, and efﬁcacy of a novel multidrug intravesical regimen consisting of Cabazitaxel, Gemcitabine, and Cisplatin (CGC) in the treatment of BCG resistant non-muscle invasive urothelial carcinoma of the bladder. This phase I trial will have a combined dose and cycle-escalation scheme with enrollment of up to 24 patients.

DETAILED DESCRIPTION:
Nonsurgical treatment strategies for BCG refractory bladder cancer have failed to prove themselves as reliable options for increased survival among this subset of bladder cancer patients. For these patients, removal of the bladder with all the associated perioperative risks and the subsequent reduction of quality of life, remains the only option. Prior attempts at second line treatments have included intravesical (within the bladder) monotherapy with a range of drugs including Gemcitabine and Paclitaxel (a taxane, similar to Cabazitaxel). These drugs have shown some potential improvement for a small number of patients Given the synergy of systemic chemotherapy, it is believed that a multidrug regimen would allow for further improvement in survival among these patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a histologically confirmed diagnosis of non- muscle invasive urothelial carcinoma of the bladder at the study institution prior to the beginning of the study. This includes patients with:

* High grade Ta papillary lesion(s)
* High or low grade T1 papillary lesion(s)
* Carcinoma In Situ (CIS), with or without Ta or T1 papillary tumor(s) of any grade The patient must have Bacillus Calmette-Guerin (BCG) refractory or recurrent non-muscle invasive bladder cancer
* Refractory disease is defined as evidence of persistent high risk bladder cancer (high grade Ta, T1 and/or CIS) at the first cystoscopic exam after the initial 6 week induction course of BCG or at the 6 month cystoscopic exam.
* Recurrent disease is defined as reappearance of disease after achieving a tumor- free status by 6 months following a full induction course of BCG with or without maintenance BCG. Participants must have recurred within 18 months following the last dose of BCG.

  * Low-grade superficial (Ta) disease will not be considered recurrent.
  * Patients must exhibit disease recurrence after receiving some form of standard intravesical therapy that must include a minimum of one induction course of BCG and may also include prior exposure to mitomycin, interferon, single agent gemcitabine or taxane therapy or maintenance.
* Patients must be eligible for radical cystectomy and refuse this standard of care treatment or not be a surgical candidate for radical cystectomy based on other comorbidities.
* All grossly visible disease in the bladder must be fully resected and pathologic stage will be confirmed at the study institution.
* Patients enrolled in other clinical trials must have received their last treatment at least 6 weeks prior to enrollment.
* Age > 18 and must be able to read, understand and sign informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance Status: ECOG of 0 or 1 including patients who are not surgical candidates due to comorbid conditions.
* Women of childbearing potential must have a negative pregnancy test.
* All patients of childbearing potential must be willing to consent to using effective contraception, i.e., intrauterine device (IUD), Birth control pills, Depo-Provera, and condoms while on treatment and for 3 months after their participation in the study ends.
* No experimental intravesical therapy within 6 weeks of study entry

Exclusion Criteria:

* History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on I these treatments)
* Concurrent malignancy diagnosed within 6 months of entry to the study.
* Concurrent treatment with any systemic chemotherapeutic agent.
* Inadequate organ and bone marrow function as evidenced by:

  * Hemoglobin: less than 8.0 g/dL
  * Absolute neutrophil count: less than 1.5 x 10^9/L
  * Platelet count: less than 80x 10^9/L
  * Aspartate Aminotransferase Test (AST) / Serum Glutamic Oxaloacetic Transaminase (SGOT) and/or ( Alanine Aminotransferase Test (ALT)/ Serum Glutamic Pyruvic Transaminase (SGPT) >2.5 x upper limit of normal (ULN);
  * Total bilirubin >1.5 x ULN
  * Serum creatinine >2 x ULN. If creatinine 1.5 - 2.0 x ULN, creatinine clearance will be calculated according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula and patients with creatinine clearance <30 mL/min should be excluded.
* Women who are pregnant or lactating.
* Documented history of vesicoureteral reflux or an indwelling urinary stent.
* Participation in any other research protocol involving administration of an investigational agent within 6 weeks prior to study entry.
* No Institutional Review Board (IRB) approved signed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1a/1b: The number of serious adverse events associated with therapy of intravesically administered Cabazitaxel, Gemcitabine, and Cisplatin. | 6 weeks from baseline
  The investigator is measuring safety by looking at the number of events that occur during the study
Phase 2: The number of complete responders after completion of six weeks of intravesically | 6 weeks from baseline
  The investigator is measuring efficacy by the number of complete responders to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guarionex DeCastro, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center - HIP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Columbia University current clinical trials — https://cancer.columbia.edu/